CLINICAL TRIAL: NCT05292807
Title: Imagery Rescripting and Imaginal Exposure for Anxiety Symptoms: Mechanisms and Outcomes in a Large Analog Sample
Brief Title: Imagery Rescripting and Imaginal Exposure for Anxiety Symptoms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebrew University of Jerusalem (Other)
Responsible Party: Principal Investigator, Jonathan D. Huppert, Professor, Hebrew University of Jerusalem
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: isf2157/2021
Record Dates: First submitted 2022-03-14; First posted 2022-03-23 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Social Anxiety; Generalized Anxiety; Obsessive-Compulsive Symptom; Panic
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Imaginal exposure for memories (Experimental): A behavioral intervention in imagery for memories
  Interventions: Behavioral: Imaginal exposure for memories
- Imaginal exposure for future events (Experimental): A behavioral intervention in imagery for future events
  Interventions: Behavioral: Imaginal exposure for future events
- Imagery rescripting for memories (Experimental): A different behavioral intervention in imagery for memories
  Interventions: Behavioral: Imagery rescripting for memories
- Imagery rescripting for future events (Experimental): A different behavioral intervention in imagery for future events
  Interventions: Behavioral: Imagery rescripting for future events

INTERVENTIONS:
Behavioral: Imaginal exposure for memories — Participants in this arm will be asked to decide alongside with the intervention provider (a clinical PhD student or M.A student under the supervision of the principal investigator) to imagine a script based on a past distressing anxiety provoking scenario multiple times while honing in on the most negative aspects.
  Arms: Imaginal exposure for memories
Behavioral: Imaginal exposure for future events — Participants in this arm will be asked to decide alongside with the intervention provider (a clinical PhD student or M.A student under the supervision of the principal investigator) to imagine a script based on a future distressing anxiety provoking scenario multiple times while honing in on the most negative aspects.
  Arms: Imaginal exposure for future events
Behavioral: Imagery rescripting for memories — Participants in this arm will be asked to decide alongside with the intervention provider (a clinical PhD student or M.A student under the supervision of the principal investigator) to imagine a script based on a past distressing anxiety provoking scenarios one time while honing in on the most negative aspects. Afterwards they will insert changes into the script that try to help them cope in the imagery: First imagining the scenario from a different character perspective that enacts changes in the memories. Second, The will imagine the scenario again from the original perspective along with changes done by the additional character.
  Arms: Imagery rescripting for memories
Behavioral: Imagery rescripting for future events — Participants in this arm will be asked to decide alongside with the intervention provider (a clinical PhD student or M.A student under the supervision of the principal investigator) to imagine a script based on a future distressing anxiety provoking scenarios one time while honing in on the most negative aspects. Afterwards they will insert changes into the script that try to help them cope in the imagery: First imagining the scenario from a different character perspective that enacts changes in the memories. Second, The will imagine the scenario again from the original perspective along with changes done by the additional character.
  Arms: Imagery rescripting for future events

SUMMARY:
This study will recruit 460 participants who self-report high symptoms of anxiety. Participants will be randomly assigned to one of 4 groups: one analog intervention of Imagery Rescripting (IR) for memories, an analog intervention of IR for future events, and analog intervention of Imaginal Exposure (IE) for memories and an analog intervention of IE for future events. We will examine the efficacy and mechanisms behind each intervention.

DETAILED DESCRIPTION:
After being informed about the study potential risks, all patients giving written informed consent will undergo screening to determine eligibility for study entry. They will be randomly assigned to one of four conditions (Imagery rescripting past; Imagery rescripting future; Imaginal exposure past; Imaginal exposure future) at a 1:1:1:1 ratio (n = 115 per group). Participant will be assigned using a variance minimization method that controls for between group variance in continuous and categorical variables- SPIN, ASI-3, OCI-R, GAD-7 and gender with a completely random assignment p random = .2 (for algorithm see Sella et al., 2018). Participants will attend three ~1.5 hour online ZOOM sessions (baseline-assessment and measurement, intervention, post assessment and measurement and follow-up measurement).

In this multiple baseline study, participant will enter the intervention phase either 7 or 14 days after the baseline stage.

Assessors will be blind to the treatment condition.

ELIGIBILITY:
Inclusion Criteria:

We will recruit participants based on attainment of SPIN score >= 24 and/or ASI-3 scores >=23 and/or OCI-R subscale scores (not including hoarding subscale) >=6 and/or GAD-7 scores >= 9 .

Exclusion Criteria:

Diagnosis of psychosis, active suicidality, post-traumatic stress disorder, acute stress disorder. Can't report a negative imagery related to a future social scenario. Attending active psychotherapy sessions. Started/stopped taking psychotherapeutic medications in the last 3 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2022-04-14 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the Social phobia inventory (SPIN) | Will be measured at Baseline (7 or 14 days before the intervention), Intervention (immediately after the intervention), post-intervention ( 7 days after the intervention) and Follow-up (28 days after the intervention)
  The SPIN is a 17-item validated self-report instrument assessing sum of social phobia symptom intensity over the past week. Possible scores range from 0 (not at all) to 4 (Extremely).
  Sum scores range is 0-68.
  Change = 1: (post-intervention score - Baseline Score) 2: (Follow-up score - Baseline Score)
Change from baseline in the Anxiety Sensitivity Index - 3 (ASI-3) | Will be measured at Baseline (7 or 14 days before the intervention), Intervention (immediately after the intervention), post-intervention (7 days after the intervention) and Follow-up (28 days after the intervention)
  The ASI-3 is an 18-item validated self-report instrument assessing sum of anxiety sensitivity symptom intensity over the past week. Possible scores range from 0 (not at all) to 4 (Very Much).
  Sum scores range is 0-72.
  Change = 1: (post-intervention score - Baseline Score) 2: (Follow-up score - Baseline Score)
Change from baseline in the Obsessive-Compulsive Inventory Revised (OCI-R) | Will be measured at Baseline (7 or 14 days before the intervention), Intervention (immediately after the intervention), post-intervention (7 days after the intervention) and Follow-up (28 days after the intervention)
  The OCI-R is an 18-item validated self-report instrument assessing sum of obsessive-compulsive symptom intensity over the past week (Taylor et al., 2007). Possible scores range from 0 (not at all) to 4 (Extremely).
  Sum scores range is 0-72.
  Change = 1: (post-intervention score - Baseline Score) 2: (Follow-up score - Baseline Score)
Change from baseline in the Generalized Anxiety Scale-7 (GAD-7) | Will be measured at Baseline (7 or 14 days before the intervention), Intervention (immediately after the intervention), post-intervention (7 days after the intervention) and Follow-up (28 days after the intervention)
  The GAD-7 is a 7-item validated self-report instrument assessing sum of generalized anxiety symptom intensity over the past week. Possible scores range from 0 (not at all) to 3 (Almost every day).
  Sum scores range is 0-21.
  Change = 1: (post-intervention score - Baseline Score) 2: (Follow-up score - Baseline Score)
Change from baseline in The Overall Anxiety Severity and Impairment Scale (OASIS) | Will be measured at Baseline (7 or 14 days before the intervention), Intervention (immediately after the intervention), post-intervention (7 days after the intervention) and Follow-up (28 days after the intervention)
  The OASIS is a 5-item validated self-report instrument assessing sum of anxiety related symptoms, distress avoidance and functioning symptom intensity over the past week (Taylor et al., 2007). Possible scores range from 0 to 4.
  Sum scores range is 0-20.
  Change = 1: (post-intervention score - Baseline Score) 2: (Follow-up score - Baseline Score)

SECONDARY OUTCOMES:
Change from Baseline in the Thought fusion inventory (TFI) | Will be measured at Baseline (7 or 14 days before the intervention), Intervention (immediately after the intervention), post-intervention ( 7 days after the intervention) and Follow-up (28 days after the intervention)
  The TFI is a validated 14 item self-reported instrument assessing average belief in statement that describe the effects of thoughts on reality, objects and actions. Possible scores range from 0 (Do not believe at all) to 100 (completely convinced it is true) in intervals of 10.
  Average score (0- 100) Change = 1: (post-intervention score - Baseline Score) 2: (Follow-up score - Baseline Score)
Change from Baseline in the Thought Action Fusion scale - Revised (TAFS-R) | Will be measured at Baseline (7 or 14 days before the intervention), Intervention (immediately after the intervention), post-intervention (7 days after the intervention) and Follow-up (28 days after the intervention)
  The TAFS-R is a validated 19 item self-reported instrument assessing belief in statement that describe the irrational assumption that just because a "bad" thought presents itself to the mind, then it is undeniably followed or accompanied by a specific "bad" action. Possible scores range from 0 (Do not agree) to 4 (Agree alot).
  Sum score (0- 76) Change = 1: (post-intervention score - Baseline Score) 2: (Follow-up score - Baseline Score)
Change from Baseline to follow-up in the amount of negative and positive/neutral content details of the memory/future imagery | Time Frame: Will be measured at Baseline (7 or 14 days before the intervention) and post-intervention ( 7 days after the intervention)
  The Waterloo Image and Memories Interview (WIMI) is a validated structured interview for assessing content of imagery and memories. valence of the details will be scored using a trained coder.
  change = post-intervention - Baseline Score. The participant provides descriptions of a negative imagery and memory related to his primary symptoms dimension.
The believability of the negative core-beliefs that the participant link to the negative imagery and memory provided in the WIMI | Time Frame: Will be measured at Baseline (7 or 14 days before the intervention) and post-intervention ( 7 days after the intervention)
  The Waterloo Image and Memories Interview (WIMI) is a validated structured interview for assessing content of core beliefs related to the future imagery and memory.
  Believability will be given by the participant for each identified core-belief on a scale of 0 (Do not believe it at all) to 100 (Completely Believe it).
  change = post-intervention - Baseline Score.
imaginal Based Approach Test (iBAT) that measures the participant's willingness to interact with pre-scripted distressing scenarios in imagination | Time Frame: Will be measured at Baseline (7 or 14 days before the intervention) and post-intervention ( 7 days after the intervention)
  The iBAT is currently being developed in our lab. The more levels the participants pass (listen to imaginal scenario in full without pressing "skip") the higher the score he receive (from 0 to 10)
  There are two versions in the task, each with different 10 scenarios. The versions will be counterbalanced across participants.
  Recruitment is completed for the first sample and pre-registration is available at the open science framework website:
  change = post-intervention - Baseline Score.
  https://osf.io/bp42h/?view_only=5211617cedf94f71a4daa746e98d924a
The Brief core schema scale (BCSS) | Will be measured at Baseline (7 or 14 days before the intervention), Intervention (immediately after the intervention), post-intervention (7 days after the intervention) and Follow-up (28 days after the intervention)
  the BCSS measures participants' self-beliefs about themselves and others. It is a well validated self-report instrument. It has 24 items total. Each item is scored from 1 (believe it slightly) to 3 (believe it totally)
  Two sum scores: self (0- 36), other (0-36) Change = 1: (post-intervention score - Baseline Score) 2: (Follow-up score - Baseline Score)
The Self compassion scale short (SCS) | Will be measured at Baseline (7 or 14 days before the intervention), Intervention (immediately after the intervention), post-intervention (7 days after the intervention) and Follow-up (28 days after the intervention)
  The SCS is a validated self-report measure, that measures participants' tendency to react to one own suffering and misfortune with self-compassion. It has 12 items with scores ranging from 1 (Almost never) to 5 (Almost always).
  Sum score (12- 60) Change = 1: (post-intervention score - Baseline Score) 2: (Follow-up score - Baseline Score)
The impact of future events scale (IFES) | Will be measured at Baseline (7 or 14 days before the intervention), Intervention (immediately after the intervention), post-intervention ( 7 days after the intervention) and Follow-up (28 days after the intervention)
  The IFES is a validated self-report measure, that measures participants' symptoms in reaction to negative future events. It has 24 items with scores ranging from 0 (Not at all) to 4 (A lot).
  Sum score (0- 96) Change = 1: (post-intervention score - Baseline Score) 2: (Follow-up score - Baseline Score)
The impact of events scale (IES) | Will be measured at Baseline (7 or 14 days before the intervention), Intervention (immediately after the intervention), post-intervention ( 7 days after the intervention) and Follow-up (28 days after the intervention)
  The IES is a validated self-report measure, that measures participants' symptoms in reaction to negative past events. It has 22 items with scores ranging from 0 (Not at all) to 4 (A lot).
  Sum score (0- 88) Change = 1: (post-intervention score - Baseline Score) 2: (Follow-up score - Baseline Score)
The distress tolerance scale (DTS) | Will be measured at Baseline (7 or 14 days before the intervention), Intervention (immediately after the intervention), post-intervention ( 7 days after the intervention) and Follow-up (28 days after the intervention)
  The DTS is a validated self-report measure, that measures participants' ability to tolerate distress. It has 15 items with scores ranging from 1 (Completely agree) to 5 (Completely do not agree).
  Sum score (15- 75) Change = 1: (post-intervention score - Baseline Score) 2: (Follow-up score - Baseline Score)
The experiences in close relationship scale short form (ECR-S) | Will be measured at Baseline (7 or 14 days before the intervention), Intervention (immediately after the intervention), post-intervention ( 7 days after the intervention) and Follow-up (28 days after the intervention)
  The ECR-S is a validated self-report measure, that measures participants' behavior in close relationships and maps these behaviors on dimensions of anxious attachment and avoidant attachment. It has 12 items with scores ranging from 1 (Strongly Disagree) to 7 (Strongly Agree).
  Two average scores: anxious attachment (1-7), other (1-7) Change = 1: (post-intervention score - Baseline Score) 2: (Follow-up score - Baseline Score)
The short form of the metacognitions questionnaire (MCQ-30) | Will be measured at Baseline (7 or 14 days before the intervention), Intervention (immediately after the intervention), post-intervention ( 7 days after the intervention) and Follow-up (28 days after the intervention)
  The MCQ-30 is a validated self-report measure, that measures participants' beliefs about their cognitions. It has 30 items with scores ranging from 1 (Do not agree) to 4 (Agree a lot).
  Sum score (30- 120) Change = 1: (post-intervention score - Baseline Score) 2: (Follow-up score - Baseline Score)
The Beck cognitive insight scale (BCIS) | Will be measured at Baseline (7 or 14 days before the intervention) and post-intervention ( 7 days after the intervention)
  The BCIS is a validated self-report measure, that measures participants' cognitive insight about their symptoms. It has 15 items with scores ranging from 0 (Do not agree) to 3 (Completely Agree).
  Sum score (0- 45) Change = 1: (post-intervention score - Baseline Score)
Locus of control scale (LOC) | Will be measured at Baseline (7 or 14 days before the intervention) and post-intervention ( 7 days after the intervention)
  The Locus of control scale measures participants feeling of control over their problems in life. It has 5 items with scores ranging from 1 (Completely not agree) to 5 (Completely Agree).
  Sum score (5- 25) Change = 1: (post-intervention score - Baseline Score)
Self-Appraisal of Illness Questionnaire (SAIQ) | Will be measured right before the Intervention, right immediately after the intervention, post-intervention ( 7 days after the intervention)
  The SAIQ assess attitudes toward mental illness among persons receiving psychiatric treatment.
  There will be 8 items from that questionnaire:
  0 (Not at all) to 3 (A great deal) In general, how much do you tend to worry? How much do you worry about your condition? How much do you worry about losing friends because of your condition? How much do you worry about being unable to work because of your condition?
  0 (Strongly agree) to 3 (Strongly Disagree) Do you believe the current treatment to be necessary? I think my condition requires psychiatric treatment I think my condition will go away by itself? If I were to discontinue treatment today I would do fine
  Change = 1: (post-intervention score - before intervention) 2: (after intervention - before intervention)
Questionnaire implicit association task (qIAT) | Time Frame: Will be measured at Baseline (7 or 14 days before the intervention) and post-intervention ( 7 days after the intervention)
  In this task, participant will classify sentences into two categories (TRUE of FALSE). Sentences are statement taken from the brief core schema scale describing self-beliefs in a positive or negative way. Participants in one block would have to respond TRUE to the positive statements and FALSE to the negative statements. In the second block, the instruction will be reversed, and participants will respond TRUE to the negative statements and FALSE to the positive statements.
  For each participant a d score will be calculated based on the algorithm in Greenwald, Nosek and Banaji (2003) paper.
  change = post-intervention - Baseline Score.
Paced visual serial addition test (PASAT) | Time Frame: Will be measured at Baseline (7 or 14 days before the intervention) and post-intervention ( 7 days after the intervention)
  The task requires participants to perform serial additions using the two previously displayed single digits (1-9) in a long running series of digits. They need to add the digits by pressing numbers presented on a circle on screen (2-18). The latency between digits begins at 3s in the initial 3 min block allowing participants to acclimatize to the task itself. The second block is 5-min long with a shorter display latency of 2 s between digits. The third block has a latency of 1s and can last for a maximum of 10 min; however, participants are instructed during the rest period that due to the difficulty they are allowed to end this block at any time by pressing a designated key on the terminals' keyboard. Duration of the third block provides a time measure for resistance to psychological stress
  change = post-intervention - Baseline Score.
Daily symptoms | [Time Frame: Daily, from Baseline to post-intervention (a total of 14, or 21 days)]
  The first 3 OASIS (see above) items pertaining to frequency, severity and avoidance of anxiety.
  Two of the following symptom focus area (based on the results from the DIAMOND interview in the baseline assessment):
  social anxiety (1-7): I was afraid I will say or do the wrong things. I was afraid what other people would think of me. I was afraid others would not accept me. Obsessions and compulsions: three items from the OCI-R that participant scored the highest at. (0-4) Anxiety sensitivity: (0-4) I was anxious that a panic attack would occur. I was anxious I would not be able to handle the panic attack. I was anxious something horrible would happen if a panic attack would occur. I tried to avoid experiencing a panic attack. Generalized anxiety: (0-4) I couldn't worrying or controlling my worry. I was so restless I had trouble sitting down without moving. I was way too worried about different things.
Daily mechanisms | [Time Frame: Daily, from Baseline to post-intervention (a total of 14, or 21 days)]
  Participants will fill out 9 items pertaining to specific symptoms and mechanisms (Not at all 0 to 100 Very much VAS):
  I believed that if I thought or imagined an unpleasant event it causes it more likely to happen.
  I believed that if I thought or imagined I would behave in a negative way it is more likely that I would actually behave this way I believed my thoughts become reality, if I think something it will come true I felt vulnerable I felt weak I tried being understanding and patient towards the aspects in my personality I do not love I try to remind myself that feelings of inadequacy are shared by most people I couldn't handle feelings of stress or distress I did everything to stop feeling stress or distress.

OTHER OUTCOMES:
Diagnostic Interview for Anxiety, Mood, and OCD and Related Neuropsychiatric Disorders (DIAMOND) | Baseline only
  This interview is based on DSM-5 (Diagnostic and Statistical Manual of Mental Disorders fifth edition) diagnostic criteria. It will allow us to detect the presence of social anxiety disorder, generalized anxiety disorder, obsessive-compulsive disorder and/or panic disorder before the start of the intervention.
  This interview will be used to exclude participants based on suicidality, psychosis, post-traumatic stress disorder, acute-stress disorder and substance abuse disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan D Huppert, PhD, Principal Investigator — Professor in the Hebrew University of Jerusalem psychology department
Locations (1):
- Hebrew University of Jerusalem, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Connor KM, Davidson JR, Churchill LE, Sherwood A, Foa E, Weisler RH. Psychometric properties of the Social Phobia Inventory (SPIN). New self-rating scale. Br J Psychiatry. 2000 Apr;176:379-86. doi: 10.1192/bjp.176.4.379. PMID 10827888
- [Background] Moscovitch DA, Vidovic V, Lenton-Brym AP, Dupasquier JR, Barber KC, Hudd T, Zabara N, Romano M. Autobiographical memory retrieval and appraisal in social anxiety disorder. Behav Res Ther. 2018 Aug;107:106-116. doi: 10.1016/j.brat.2018.06.008. Epub 2018 Jun 22. PMID 29960125
- [Background] Tolin DF, Gilliam C, Wootton BM, Bowe W, Bragdon LB, Davis E, Hannan SE, Steinman SA, Worden B, Hallion LS. Psychometric Properties of a Structured Diagnostic Interview for DSM-5 Anxiety, Mood, and Obsessive-Compulsive and Related Disorders. Assessment. 2018 Jan;25(1):3-13. doi: 10.1177/1073191116638410. Epub 2016 Mar 17. PMID 26988404
- [Background] Meyer JF, Brown TA. Psychometric evaluation of the thought-action fusion scale in a large clinical sample. Assessment. 2013 Dec;20(6):764-75. doi: 10.1177/1073191112436670. Epub 2012 Feb 6. PMID 22315482
- [Background] Foa EB, Huppert JD, Leiberg S, Langner R, Kichic R, Hajcak G, Salkovskis PM. The Obsessive-Compulsive Inventory: development and validation of a short version. Psychol Assess. 2002 Dec;14(4):485-96. PMID 12501574
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Deeprose C, Malik A, Holmes EA. Measuring Intrusive Prospective Imagery using the Impact of Future Events Scale (IFES): Psychometric properties and relation to risk for Bipolar Disorder. Int J Cogn Ther. 2011 Jun;4(2):187-196. doi: 10.1521/ijct.2011.4.2.187. PMID 22984633
- [Background] Strachan LP, Hyett MP, McEvoy PM. Imagery Rescripting for Anxiety Disorders and Obsessive-Compulsive Disorder: Recent Advances and Future Directions. Curr Psychiatry Rep. 2020 Feb 19;22(4):17. doi: 10.1007/s11920-020-1139-4. PMID 32076845
- [Background] van Minnen A, Foa EB. The effect of imaginal exposure length on outcome of treatment for PTSD. J Trauma Stress. 2006 Aug;19(4):427-38. doi: 10.1002/jts.20146. PMID 16929519
- [Background] Garner LE, Van Kirk N, Tifft ED, Krompinger JW, Mathes BM, Fraire M, Falkenstein MJ, Brennan BP, Crosby JM, Elias JA. Validation of the distress tolerance scale-short form in obsessive compulsive disorder. J Clin Psychol. 2018 Jun;74(6):916-925. doi: 10.1002/jclp.22554. Epub 2017 Nov 15. PMID 29139125
- [Background] Raes F, Pommier E, Neff KD, Van Gucht D. Construction and factorial validation of a short form of the Self-Compassion Scale. Clin Psychol Psychother. 2011 May-Jun;18(3):250-5. doi: 10.1002/cpp.702. Epub 2010 Jun 8. PMID 21584907
- [Background] Pedersen G, Eikenaes I, Urnes O, Skulberg GM, Wilberg T. Experiences in Close Relationships - Psychometric properties among patients with personality disorders. Personal Ment Health. 2015 Aug;9(3):208-19. doi: 10.1002/pmh.1298. Epub 2015 Jun 1. PMID 26033784
- [Background] Campbell-Sills L, Norman SB, Craske MG, Sullivan G, Lang AJ, Chavira DA, Bystritsky A, Sherbourne C, Roy-Byrne P, Stein MB. Validation of a brief measure of anxiety-related severity and impairment: the Overall Anxiety Severity and Impairment Scale (OASIS). J Affect Disord. 2009 Jan;112(1-3):92-101. doi: 10.1016/j.jad.2008.03.014. Epub 2008 May 16. PMID 18486238
- [Background] Faustino B. Maladaptive and Adaptive Cognitions About the Self and Others: Confirmatory Factor Analysis of the Brief Core Schemas Scales. Psychol Rep. 2023 Jun;126(3):1445-1460. doi: 10.1177/00332941211063602. Epub 2022 Jan 11. PMID 35015611
- [Background] Horowitz M, Wilner N, Alvarez W. Impact of Event Scale: a measure of subjective stress. Psychosom Med. 1979 May;41(3):209-18. doi: 10.1097/00006842-197905000-00004. PMID 472086
- [Background] Greenwald AG, Nosek BA, Banaji MR. Understanding and using the implicit association test: I. An improved scoring algorithm. J Pers Soc Psychol. 2003 Aug;85(2):197-216. doi: 10.1037/0022-3514.85.2.197. PMID 12916565
- [Background] Ozakbas S, Cinar BP, Gurkan MA, Ozturk O, Oz D, Kursun BB. Paced auditory serial addition test: National normative data. Clin Neurol Neurosurg. 2016 Jan;140:97-9. doi: 10.1016/j.clineuro.2015.11.014. Epub 2015 Nov 24. PMID 26688504
- [Background] Sella F, Raz G, Cohen Kadosh R. When randomisation is not good enough: Matching groups in intervention studies. Psychon Bull Rev. 2021 Dec;28(6):2085-2093. doi: 10.3758/s13423-021-01970-5. Epub 2021 Jul 9. PMID 34244982